CLINICAL TRIAL: NCT06898190
Title: Testing the Feasibility & Fidelity of the Learning Early Infant Feeding Cues (LEIFc) Intervention
Brief Title: Testing LEIFc in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jessica Bahorski, Associate Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002895
Record Dates: First submitted 2025-03-16; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Responsive Infant Feeding; Infant Growth
Keywords: infants; infant feeding; breastfeeding; health promotion; infant growth; childhood obesity prevention
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Obesity-Related Behavioral Intervention Trials (ORBIT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LEIFc (Experimental): The LEIFc intervention was developed by the research team and includes several key components, including a prenatal visit to introduce infants' early feeding cues and in the moment coaching supports during feeding routines after the baby is born. The SS-OO-PP-RR ("super," Setting the Stage, Observation and Opportunities, Problem Solving and Planning, Reflection and Review) coaching approach is a hallmark of the intervention that is intended to build caregiver confidence in reading their child's cues with in the moment practice and feedback as well as problem solving and reflecting on what is working or what needs to be adapted.
  Interventions: Behavioral: Learning Early Infant Feeding Cues (LEIFc)

INTERVENTIONS:
Behavioral: Learning Early Infant Feeding Cues (LEIFc) — Coaching sessions using SS-OO-PP-RR are conducted at infant age of 2 and 3 months. This occurs during an infant feeding session between mother and infant with the interventionists offering coaching specific to responsive feeding during the session. At the conclusion of the visit, the interventionists and mother develop specific strategies to practices prior to the next visit. At the following visit, a discussion of reflection and review occurs prior to the infant feeding session to identify what is going well and what still needs work.

SUMMARY:
The reason that we are doing this research is to teach mothers ways to communicate with their baby during feeding. Understanding signals a baby gives helps mothers know when and how much to feed their baby which will help the baby grow in a healthy way.

There are 5 study visits, 1 during pregnancy and 4 after the baby is born. At the first visit participants will watch some videos about feeding babies and be provided with information to read about feeding babies, there is also a questionnaire to complete. After the baby is born, a research team member will come to participants' homes at infant age of 1, 2, 3, and 4 months to videotape an infant feeding session. At the visit when the baby is 2 and 3 months of age, the intervention will occur in which the interventionists will provide coaching about responsive feeding before and during a feeding session. The baby's height and weight will be collected and some questionnaires completed. At the last study visit, a research assistant will ask opened ended questions about the study itself, these questions and participant answers will be audio recorded.

DETAILED DESCRIPTION:
3.0 Background* 3.1 and 3.3 Health disparities in pediatric obesity are staggering; Non-Hispanic black and Hispanic children have obesity rates (22.2% and 25.8% respectively) higher than the national average (18.5%) and higher than non-Hispanic white children (14.1%).1,2 Additionally, children of low socioeconomic status (SES) are more likely to have obesity.2,3 These same populations are disproportionately affected by lifelong cardiometabolic conditions that result from obesity such as hypercholesterolemia, hypertension, and type 2 diabetes.4 Children with obesity are also more likely to suffer from mental health disorders (i.e., depression, anxiety) and complications of the pulmonary, orthopedic, and gastrointestinal systems.2,5,6 Lifestyle modifications implemented early in life are key to preventing obesity and the resulting lifelong complications. The first 1,000 days of life, from conception to age two years, is a critical period for development of habits that contribute to one's weight status later in life, such as dietary preferences and behaviors.7-10 Therefore, interventions implemented during the first 1,000 days and targeting infants from high-risk groups have potential to decrease one's obesity risk and address racial/ethnic and socioeconomic health disparities.

Infant feeding practices, which include what and how infants are fed, are one such habit that could be modified to decrease obesity risk.5 Exclusive formula feeding, short duration of breastfeeding when initiated, and early introduction of complementary foods contribute to rapid infant weight gain which, in turn, contributes to higher risk for childhood obesity.11,12 Many initiatives have targeted "what" infants are fed (i.e., promoting breastfeeding and healthy dietary intake) whereas "how" infants are fed is also important, yet understudied.5,8,13,14 The responsive feeding approach is thought to promote the ability to recognize and respond to internal cues of hunger and satiety.13-17 The ability to recognize these internal cues and self-regulate intake in response to physiologic need is associated with healthy weight gain trajectories.13,16 Responsive feeding occurs when a parent (or other caregiver) learns and recognizes the infant's cues of hunger and satiety, and responds promptly to these cues.18 The Dietary Guidelines for Americans recommend responsive feeding.19 Additionally, a recent systematic review found responsive feeding to be associated with healthy growth in children less than two years of age.13 Education on, and promotion of, responsive feeding should begin prenatally and evolve with the development of the child.18 Infant feeding during the first months after birth often occurs in the home, making this an ideal environment to promote responsive feeding.10,20-22 Interventions to promote responsive feeding have shown benefit in preventing rapid infant weight gain and promoting healthy dietary patterns in young children.20-28 However, this research has not been integrated using a validated coaching approach with the family's home. Additionally, responsive feeding has been largely measured via surveys.25 To address these gaps, an individualized responsive feeding coaching intervention, Learning Early Infant Feeding Cues (LEIFc), has been developed by the PI of the proposed study and her team.

The multicomponent LEIFc intervention involves maternal education on responsive feeding practices while using a family-guided caregiver coaching approach called SS-OO-PP-RR (Setting the Stage, Observation and Opportunities, Problem Solving and Planning, Reflection and Review) during feeding sessions.29,30 The SS-OO-PP-RR approach was developed based on adult learning theory and has been successfully used with parents and childcare providers to promote development across domains in infants and young children.29-31 For the LEIFc intervention, SS-OO-PP-RR was modified to be specific to communication during feeding to promote responsive feeding (Table 1). It is used as a guide for the interventionists during the coaching session but will also be used to evaluate the fidelity of the intervention. The purpose of this study is to test fidelity and feasibility of the LEIFc intervention in a group of diverse mother-infant dyads North Florida.

4.0 Study Endpoints* 4.1 The study will end when the participants complete all time points or the infant reaches 6 months of age.

5.0 Study Intervention

1.1 The investigators developed the LEIFc intervention based on the literature and prior pilot studies. The multicomponent LEIFc intervention involves maternal education on responsive feeding practices while using a family-guided caregiver coaching approach called SS-OO-PP-RR (Setting the Stage, Observation and Opportunities, Problem Solving and Planning, Reflection and Review) during feeding sessions.29,30 The SS-OO-PP-RR approach was developed based on the adult learning theory and has been successfully used with parents and childcare providers to promote development across domains in infants and young children.29-31 For the LEIFc intervention, SS-OO-PP-RR was modified to be specific to communication during feeding to promote responsive feeding. It is used as a guide for interventionists during the coaching session but will also be used to evaluate the fidelity of the intervention. The research study consists of five visits (Table 1) beginning in the third trimester (28 weeks and beyond) of pregnancy to four months after the infant's birth.

6.0 Procedures Involved* Design. This study uses a pre-post quasi experimental design with no control group to examine the feasibility, utility, and social validity of the LEIFc intervention. Videos will be coded prior to the intervention then after two coaching sessions between interventionist and mother during a feeding session. We will also use a pre-post measure to assess mother knowledge and beliefs regarding infant feeding practices. Demographic factors, post-partum depression, and maternal-infant bonding will be considered as covariates.

Instruments. Objective measurement of responsive feeding will occur through video coding and analysis of feeding sessions. The research team is in the process of developing a coding scheme. The Responsiveness to Child Feeding Cues Scale (RCFCS) 32 and literature from the communication arena 33-35 have been used to guide the coding scheme. Research assistants will be trained on the coding scheme and will use existing videos to code with a goal of at least 85% agreement achieved to confirm interrater reliability. Investigator Romano has significant experience with observational measurement.

The Infant Feeding Questionnaire (IFQ) is completed by mothers and provides a measure of infant feeding practices and beliefs.36 The 20-item questionnaire assesses for: concern for the infant being underweight, concern about hunger, awareness of hunger and fullness cues, concern about overweight, feeding on a schedule, providing food to calm an infant, and social interaction during feeding.36 Likert-type scoring is used, higher scores indicate a stronger measure of the construct. Investigator Bahorski has prior experience using this tool. 37,38 Infant feeding practices, including breastmilk, formula, and/or complementary foods, are collected at each visit, as well as reflective feedback from the interventionist. This instrument was developed by the investigators based on the literature and prior research. Infant height and weight will be collected using standard clinical techniques. The Patient Health Questionnaire-9 (PHQ-9) will provide a method to screen for depression at each visit as depression is known to influence infant feeding practices.39 The Maternal-to-Infant Bonding Questionnaire (MIBQ) will be also be collected at each visit; bonding will be used as a covariate.

Procedures:

Prenatal Intervention, Phase 1 (Visit 1). Teaching about responsive feeding practices before birth. This aspect of the intervention includes written and video materials about responsive feeding practices during the mothers' final weeks of her pregnancy. These practices include hunger and satiety cues, avoiding scheduled feedings and feeding to soothe, and how to make feeding times valuable contexts for mother-infant bonding and language learning. The materials will include examples of infant cues and will engage mothers to reflect on how these practices are similar to, or different from, what she has heard about feeding from family, friends, her community, or her healthcare provider. Additionally, the mother will complete the following surveys: demographics, prenatal infant feeding plans, depression (PHQ-9), and mother-infant bonding (MIBQ). This session will be held over the phone.

Pre-test (Visit 2). Approximately two weeks after the mother's due date, participants will be contacted to confirm continued eligibility in the study (full term birth of the infant, no complications at birth or unexpected infant anomaly). If the dyad remains eligible to participate in the study, study Visit 2 will occur when the infant is approximately 1 month of age. A feeding session with mother and infant will be videotaped in the home by the interventionist (or in the clinic if the mother prefers). Surveys will include birth history, current feeding practices, IFQ, PHQ-9, and MIBQ. Infant height and weight will also be collected.

Intervention Phase 2 (Visits 3 & 4): The interventionist will conduct two study visits when the infant is approximately two and three months of age. These will be held within the family home at a time convenient to the mother (or in the clinic if the mother prefers). During these video-recorded coaching sessions, the interventionist will use a modified version of the SS-OO-PP-RR coaching approach to share the content about responsive feeding practices and responsive interactions. The mother will have a chance to practice these techniques with her infant with guidance and support from the interventionist. The mother and interventionist will also reflect and problem solve about how the interactions went and what potential adaptations could be made (i.e., if a mom is worried about wasting milk, how might they prepare bottles to account for responsiveness to a child's fullness cues). Current infant feeding practices will be collected at each visit and the PHQ-9 and MIBQ will be completed.

Post Test (Visit 5). The final visit will occur when the infant is approximately 4-5 months of age (but not more than 6 months). The interventionist will video record mother-infant interactions during a feeding as the post-test observational measure. The mother will also complete the IFQ, PHQ-9, and MIBQ; current infant feeding, infant height and weight will be collected. Maternal feedback on the intervention will be collected via open ended questions. Maternal response to questions will be audio recorded.

10.0 Subject Population* 10.1 Sample. Pregnant mothers (N = 50) aged 18 years or older, in their third trimester (28 weeks and beyond) of a healthy, singleton pregnancy will be recruited to participate in this study. Inclusion of this population of mothers will eliminate cofounding variables such as birth at either end of the age spectrum (i.e., teenage or advanced maternal age), caring for twins, or infants with complex medical conditions (i.e., congenital or genetic anomalies). Infants will be included once birth until infant age of 4-6 months. Only healthy, full-term infants with no congenital anomalies or medication conditions that would interfere with feeding and/or growth.

10.2 Women unable to provide consent will be excluded from participating along with incarcerated women.

10.3 Pregnant women and infants are included in this study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant in the 3rd trimester (28 weeks or beyond) of a healthy pregnancy
* pregnant with a single fetus
* 18 years or older
* no known complications or genetic anomalies of the infant that would interfere with feeding or growth after birth
* English or Spanish speaking

Exclusion Criteria:

* mother less than 18 years
* will not have custody of the infant after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be pregnant to be enrolled thus must be biologically female.
Enrollment: 29 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Responsive Infant Feeding | Pre-intervention (infant age 1 month) to post-intervention (infant age 4 months)
  Subjective (via survey) and objective (via video) measurement of responsive feeding will be collected pre-post intervention visits. The Infant Feeding Questionnaire will provide a subjective measure of responsive feeding. A feeding session will be video recording then coded for instances of infant cues and maternal response to cues to provide an objective measure of responsive feeding.

SECONDARY OUTCOMES:
Duration of Breastfeeding | weeks since birth
  Current infant feeding practices are collected at each study visit. Duration of any breastfeeding will be tabulated into a variable.
Age of complementary food introduction | weeks since birth
  Current infant feeding practices are collected at each study visit. The infant age (in weeks) at which any foods other than breastmilk or formula were given will be tabulated into a variable.
Infant weight-for-length z-score (WLz) | birth to 4 months
  Infant WLz will be calculated from infant weight and length measurements obtained at each study visit. The difference in WLz between infant age of 2 weeks and 6 months will be calculated. Infants will be categorized into 3 growth categories: expected growth (WLz SD change between -0.67 and 0.67, rapid growth > or equal to 0.67, or slow growth < or equal to -0.67.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD may result in a breach of confidentiality, aggregated data may be shared via a DUA.

REFERENCES:
- [Background] Bahorski J, Romano M, McDougal JM, Kiratzis E, Pocchio K, Paek I. Development of an Individualized Responsive Feeding Intervention-Learning Early Infant Feeding Cues: Protocol for a Nonrandomized Study. JMIR Res Protoc. 2023 Feb 28;12:e44329. doi: 10.2196/44329. PMID 36853761